CLINICAL TRIAL: NCT03359980
Title: Treatment of Steroid Refractory Gastro-intestinal Acute Graft-versus-Host disEase afteR AllogeneiC Hematopoietic Stem celL Transplantation With fEcal Microbiota tranSfer
Brief Title: Treatment of Steroid Refractory Gastro-intestinal Acute GVHD afteR AllogeneiC HSCT With fEcal Microbiota tranSfer
Acronym: HERACLES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPOH03
Record Dates: First submitted 2017-11-20; First posted 2017-12-02 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treated patients (Experimental): Treated with Fecal Microbiota Transfer (FMT)
  Interventions: Drug: fecal microbiota transfer

INTERVENTIONS:
Drug: fecal microbiota transfer — transfer of fecal microbiota from healthy donors to the patients
  Other Names: MaaT013

SUMMARY:
Patients who have a gastrointestinal acute Graft versus host disease (GVHD) received a first-line standard treatment of corticosteroids. For patients who do not respond or progress after an initial response have a high mortality. There is an interest in identifying effective second line therapy for these patients corticosteroid-resistant acute GVHD. Fecal microbiota transfer might be a beneficial treatment in this clinical situation with a poor prognosis and limited therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Patients who develop a first episode of Stage 2 to 4 Gastro-intestinal Acute Graft-versus-Host (GI-aGVHD) with gut predominance (Przepiorka D, 1995), resistant to a first line therapy with steroids (lack of improvement after 5 days or progression after 3 days of treatment with corticosteroids at 2 mg/Kg methylprednisolone equivalent dose) (SR GI-aGVHD)
* Age ≥ 18 years old
* Allogeneic Hematopoietic stem cell transplantation (Allo-HSCT) with any type of donor, stem cell source, GVHD prophylaxis or conditioning regimen
* Patients able to have a minimum of 12 hours discontinuation of systemic antibiotics in order to perform the allogeneic FMT
* Signature of informed and written consent by the subject or by the subject's legally acceptable representative

Exclusion Criteria:

* Grade IV hyper-acute GVHD
* Overlap chronic GVHD
* Acute GVHD after donor lymphocytes infusion
* Relapsed/persistent malignancy requiring rapid immune suppression withdrawal
* Active uncontrolled infection according to the attending physician
* Other systemic drugs than corticosteroids for GVHD treatment (including extra-corporeal photopheresis). Drugs already being used for GVHD prevention (eg. calcineurin inhibitors) are allowed.
* Absolute neutrophil count < 0.5 x 10^9 /L
* Absolute platelet count < 10 000
* Patient Epstein-Barr Virus (EBV) negative
* Evidence of toxic megacolon or gastrointestinal perforation on abdominal X-ray
* Known allergy or intolerance to trehalose or maltodextrin
* Pregnancy: positive urinary or blood test in female of childbearing potential; lactation; absence of effective contraceptive method for female of childbearing potential
* Other ongoing interventional protocol that might interfere with the current study primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Efficacy of FMT in the treatment of Steroid Refractory -Gastro-intestinal Acute GVHD (SR-GI-aGVHD) at D28 post inclusion | up to 4 weeks post inclusion
  Proportion of patients achieving GI and overall GVHD response by D28, defined as Complete response (CR) or Very Good Partial Response (VGPR)

SECONDARY OUTCOMES:
Safety of FMT in patients with SR-GI-aGVHD | through study completion, an average of six months
  The overall safety of the study will be evaluated with the incidence of all Adverse Events (AEs) and Serious Adverse Events (SAEs) (frequency, grade, relationship) throughout the study period
Gastrointestinal GVHD overall response rate at D28 post inclusion | Day 28
  Proportion of patients achieving GI and overall GVHD response by D28, defined as Complete response (CR) or Very Good Partial Response (VGPR) or Partial Response (PR)
Number of patients with infectious disorders | through study completion, an average of six months
  Evaluation of FMT activity on infectious disorders
Number of multidrug resistant bacteria in faeces | through study completion, an average of six months
  Evaluation of FMT activity on multidrug-resistant bacteria (MDRB) carriage
Number of patients with Chronic GVHD | through study completion, an average of six months
  Chronic GVHD expression

CONTACTS AND LOCATIONS:
Overall Officials: Florent Malard, MD, PhD, Principal Investigator — Hôpital Saint Antoine - PARIS
Locations (16):
- France (12):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHRU Besançon, Besançon
  - Hôpital Henri Mondor, Créteil
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Nantes, Nantes
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - CHU Strasbourg, Strasbourg
  - IUCT Oncopole, Toulouse
- Gemelli Hospital, Roma, Italy
- Poland (3):
  - Klinika Hematologii i Transplantologii, Gdansk
  - Public Clinic Hospital, Katowice
  - University Clinical hospital, Wroclaw

REFERENCES:
- [Derived] Malard F, Loschi M, Huynh A, Cluzeau T, Guenounou S, Legrand F, Magro L, Orvain C, Charbonnier A, Panz-Klapuch M, Desmier D, Mear JB, Cornillon J, Robin C, Daguindau E, Bilger K, Vehreschild MJGT, Chevallier P, Labussiere-Wallet H, Mediavilla C, Couturier MA, Bulabois CE, Camus V, Chantepie S, Ceballos P, Gaugler B, Holler E, Dore J, Prestat E, Gasc C, Plantamura E, Mohty M. Pooled allogeneic faecal microbiota MaaT013 for steroid-resistant gastrointestinal acute graft-versus-host disease: a single-arm, multicentre phase 2 trial. EClinicalMedicine. 2023 Jul 26;62:102111. doi: 10.1016/j.eclinm.2023.102111. eCollection 2023 Aug. PMID 37654670